CLINICAL TRIAL: NCT04812548
Title: A Single-arm, Open-label, Phase II Study of Sabatolimab in Combination With Azacitidine and Venetoclax in Adult Participants With High or Very High Risk Myelodysplastic Syndromes (MDS) as Per IPSS-R Criteria
Brief Title: A Study of Sabatolimab in Combination With Azacitidine and Venetoclax in High or Very High Risk MDS Participants
Acronym: STIMULUS-MDS3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped following a strategic decision from the Sponsor. It was not based on any safety findings or safety concerns with sabatolimab.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453B12203; 2020-003669-21 (EudraCT Number)
Record Dates: First submitted 2021-02-23; First posted 2021-03-23 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: MGM453; Phase II; sabatolimab; TIM-3; venetoclax; azacitidine; Myelodysplastic syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — sabatolimab; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sabatolimab + azacitidine + venetoclax (Experimental): Part 1: Safety run-in consisted of 2 subsequent cohorts of a lower dose (cohort 1) and a higher dose (cohort 2) of sabatolimab in combination with fixed dose of venetoclax and azacitidine.
  Part 2 (did not start as recruitment was stopped in Part 1) Expansion was to enroll additional participants to further investigate the regimen including sabatolimab at the higher dose, azacitidine and venetoclax. Participants data from Part 1 and Part 2 treated with the higher dose was to have been combined to determine the complete remission rate.
  Interventions: Drug: sabatolimab; Drug: azacitidine; Drug: venetoclax

INTERVENTIONS:
Drug: sabatolimab — Sabatolimab was administered at a low dose (Safety run-in (Part 1) cohort 1) or a high dose (Safety run-in (Part 1) cohort 2) via i.v. infusion over 30 minutes on Day 8 of every treatment cycle. Cycle = 28 days
  Other Names: MBG453
Drug: azacitidine — A standard dose of azacitidine was given subcutaneously or intravenously every day for seven consecutive days on days 1-7 of a confirmed treatment cycle. In keeping with standard clinical practice, the alternative schedules for five consecutive days on days 1-5, followed by a two day break, then two consecutive days on days 8-9 was permitted (alternative schedule).
Drug: venetoclax — Venetoclax film-coated tablets was administered at a dose of 400 mg orally or corresponding reduced dose for concomitant use with P-gp inhibitors or moderate or strong CYP3A4 inhibitors, once a day, from C1D1 to C1D14 during the treatment cycle. No ramp-up for venetoclax was necessary.

SUMMARY:
The purpose of the study was to find out if the new drug sabatolimab when given in combination with azacitidine and venetoclax, was safe and had beneficial effects in participants with high or very high risk myelodysplastic syndrome (MDS) who were not suitable for treatment with intensive chemotherapy or a stem-cell transplant (HSCT).

DETAILED DESCRIPTION:
Approximately 76 people with high or very high risk myelodysplastic syndrome (MDS) and age ≥ 18 years were to be asked to join this study but due to the decision by Novartis to halt recruitment the study did not enroll the approximately 76 participants.

The primary purpose of Part 1 (Safety run-in) was to rule out excessive toxicity of sabatolimab, when administered in combination with azacitidine and venetoclax. The primary purpose of the combined cohort 2 of the Safety run-in (Part 1) and Expansion (Part 2) was to have evaluated efficacy of sabatolimab, when administered in combination with azacitidine and venetoclax in adult participants with high or very high risk MDS. But due to the decision by Novartis to halt recruitment at the end of the Safety run-in, the study enrolled participants in Part 1 only.

This study was to have consisted of two parts:

Safety Run-in Part:

The first approximately 18 participants to have joined the study would have been part of the safety run-in. The first approximately 6 participants would have been enrolled to the lower dose given every four weeks sabatolimab safety run-in cohort.

After these participants would have completed 2 cycles of treatment a decision would have been made to confirm whether the chosen combination of sabatolimab with azacitidine and venetoclax was considered safe to continue with approximately 12 participants, to have been enrolled to the higher dose given every four weeks safety run-in cohort. After these participants would have completed 2 cycles of treatment a decision would have been made to confirm whether the chosen combination of sabatolimab with azacitidine and venetoclax was considered safe to continue with expansion part of the study.

Expansion Part (which did not occur):

After the safety run-in part would have confirmed that the study treatment (higher dose of sabatolimab given every four weeks with azacitidine and venetoclax) was safe, about 58 more participants would have been enrolled in the expansion part to better investigate the efficacy of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Age ≥ 18 years at the date of signing the informed consent form (ICF)
3. Morphologically confirmed diagnosis of myelodysplastic syndrome (MDS) based on 2016 WHO classification (Arber et al, 2016) by local investigator assessment with one of the following Prognostic Risk Categories, based on the revised International Prognostic Scoring System (IPSS-R) (Greenberg et al 2012):

   * Very high (> 6 points)
   * High (> 4.5-6 points)
4. Not immediately eligible for hematopoietic stem-cell transplantation (HSCT) or intensive chemotherapy at the time of screening due to individual clinical factors such as age, comorbidities and performance status, donor availability (de Witte et al 2017)
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

1. Prior exposure to TIM-3 directed therapy or any BCL-2 inhibitor (including venetoclax) at any time
2. Prior therapy with immune check point inhibitors (e.g. anti-CTLA4, anti-PD-1, anti-PD-L1, or anti-PD-L2) or cancer vaccines is not allowed if the last dose of the drug was administered within 4 months prior to start of treatment
3. Previous first-line treatment for very high risk or high risk myelodysplastic syndromes (based on IPSS-R,Greenberg et al 2012 and Arber et al, 2016) with any antineoplastic agents, approved or investigational, including for example chemotherapy, lenalidomide and hypomethylating agents (HMAs) such as decitabine or azacitidine However, a one single cycle of HMAs treatment only started prior to enrollment is allowed.
4. Live vaccine administered within 30 days prior to start of treatment
5. Current use or use within 14 days prior to start of treatment of systemic steroid therapy (> 10 mg/day prednisone or equivalent) or any immunosuppressive therapy. Topical, inhaled, nasal, ophthalmic steroids are allowed. Replacement therapy, steroids given in the context of a transfusion, are allowed and not considered a form of systemic treatment
6. History of severe hypersensitivity reactions to any ingredient of study drug(s) (azacitidine, venetoclax or sabatolimab) or monoclonal antibodies (mAbs) and/or their excipients
7. Participants with Myelodysplastic syndrome (MDS) based on 2016 WHO classification (Arber et al, 2016) with revised International Prognostic Scoring System (IPSS-R) ≤ 4.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Novartis Investigative Site, Brasschaat, Belgium
- France (2):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
- Germany (2):
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Stuttgart
- Greece (2):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Nyíregyháza, Hungary
- Novartis Investigative Site, Genova, GE, Italy
- Novartis Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten centers across 7 countries enrolled a total of 20 participants in this study.
Pre-assignment Details: Prior to dosing at Cycle 1 Day 1, participants who fulfilled all the inclusion/exclusion criteria were enrolled via IRT and a treatment number was provided for the study treatments sabatolimab, venetoclax, and azacitidine.
Groups:
- Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1): Part 1 Cohort 1: Safety run-in cohort of a lower dose of sabatolimab in combination with fixed dose of venetoclax and azacitidine.
- Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2): Part 1 Cohort 2: Safety run-in cohort of a higher dose of sabatolimab in combination with fixed dose of venetoclax and azacitidine.
Period: Overall Study
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Started | 5 | 15
Did Not Enter Post-treatment Follow-up | 1 | 5
Entered Post-treatment Follow-up | 4 | 10
Completed (Completed = completed treatment Not completed = discontinued from treatment) | 0 | 0
Not Completed | 5 | 15
Not completed — Adverse Event | 2 | 7
Not completed — HSCT Planned | 2 | 3
Not completed — Progressive Disease | 0 | 2
Not completed — Death | 0 | 1
Not completed — Post Study Access to Treatment | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS):
Groups:
- Total: Total of all reporting groups
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) | Total
Number analyzed (Participants) | 5 | 15 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (11.28) | 69.3 (9.45) | 68.8 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 5 | 11 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 14 | 18
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Dose Limiting Toxicities (DLTs) - All Grades (Safety run-in Patients Only)
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value considered by the Investigator to be at least possibly related to sabatolimab as a single contributor or in combination with other component(s) of study treatment that occurs during the DLT observation period and meets severity criteria as per protocol.
Time Frame: From Cycle 1 Day 8 to end of Cycle 2 (Cycle = 28 Days)
Population: Dose determining set (DDS): The DDS included all participants from the FAS enrolled in the Safety run-in part who met the minimum exposure criterion and had sufficient safety evaluations or experienced a dose limiting toxicity (DLT) during the first two cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 4 | 13
Participants
  Number of participants with at least one event | 0 | 2
  Blood and lymphatic system disorders (Thrombocytopenia) | 0 | 1
  Nervous system disorders (Haemorrhage intracranial) | 0 | 1

2. Primary Outcome: Percentage of Participants (Receiving 800mg Sabatolimab) Achieving Complete Remission (CR) Per Investigator Assessment
Description: This endpoint assessed Complete Remission (CR) Rate of participants from Cohort 2 of Part 1 and Part 2 according to Investigator assessment per modified IWG-MDS - Cheson 2006 criteria. CR is defined as follows: bone marrow blasts <=5%, hemoglobin level ≥ 10 g/dL, platelets count ≥ 100*10^9/L, neutrophils count ≥ 1.0*10^9/L, absence of blasts in peripheral blood.
Time Frame: up to approx. 23 months
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) comprises all participants who received at least one dose of study treatment. If a participant were assigned to a specific cohort without any administration of sabatolimab, but received venetoclax or azacitidine, the participant is included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 15
Participants | 1

3. Secondary Outcome: Percentage of Subjects Achieving a Complete Remission (CR) + Morphologic Complete Remission (mCR): Safety run-in (Part 1)
Description: Assessed the durability of complete remission (CR) or morphologic complete remission (mCR) rate. mCR is defined as <=5% blasts and blast count decrease by >=50% compared to baseline as per modified IWG-MDS Cheson 2006 criteria.
Time Frame: up to approx. 23 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 5 | 15
Participants | 4 | 13

4. Secondary Outcome: Overall Response Rate (ORR) of Participants Who Achieved Hematologic Improvement (HI) or Better as Best Response
Description: The percentage of participants achieving [CR + mCR + partial remission (PR) + hematologic improvement (HI)], per modified IWG-MDS Cheson 2006 criteria. Partial response (PR): all complete response (CR) criteria except >=50% decrease from baseline in blasts in bone marrow AND blast count in bone marrow >5%. HI (erythroid response or platelet response or neutrophil response) must last at least 8 weeks.
Time Frame: up to approx. 23 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 5 | 15
Participants | 4 | 13

5. Secondary Outcome: Percentage of Participants Who Are RBC/Platelets Transfusion Independent
Description: Improvement in red blood cells (RBC)/platelets transfusion post-baseline as per International Working Group - Myelodysplastic syndromes (IWG-MDS) by dose level for the safety run-in part (Cohort 1 (400 mg Q4W) and Cohort 2 (800 mg Q4W)) and for participants treated with sabatolimab 800 mg (Q4W) (Cohort 2 of safety run-in and expansion parts). RBC/Platelets transfusion independence is defined as participants having received no RBC/Platelets transfusions during at least 8 consecutive weeks after start of treatment.
Time Frame: up to approx. 23 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 5 | 15
Participants
  RBC | 2 | 5
  Platelets | 2 | 7

6. Secondary Outcome: Duration of Transfusion Independence
Description: Sum of each period of the transfusion independence for participants with at least one period of transfusion independence post-baseline by dose level for the safety run-in part (Cohort 1 (400 mg Q4W) and Cohort 2 (800 mg Q4W)) and for participants treated with sabatolimab 800 mg (Q4W) (Cohort 2 of safety run-in and expansion parts) for both red blood cells and platelets. RBC/Platelets transfusion independence is defined as participants having received no RBC/platelets transfusions during at least 8 consecutive weeks after start of treatment.
Time Frame: up to approx. 23 months
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) comprises all participants who received at least one dose of study treatment. If a participant were assigned to a specific cohort without any administration of sabatolimab, but received venetoclax or azacitidine, the participant is included in the analysis. Analysis is based on participants with at least one period of transfusion independence post-baseline.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 2 | 7
Weeks
  Packed Red Blood Cells: number analyzed (Participants) | 2 | 5
  Packed Red Blood Cells | 16.43 (0.808) | 23.11 (12.636)
  Platelets | 18.93 (2.727) | 24.02 (16.423)

7. Secondary Outcome: Peak Serum Concentration (Cmax) of Sabatolimab
Description: Maximal concentration of sabatolimab for participants treated with sabatolimab by dose level for the safety run-in part (Cohort 1 (400 mg Q4W) and Cohort 2 (800 mg Q4W)).
Time Frame: Continuously collected for patients during treatment with sabatolimab up to 150 days after last treatment, approx. 23 months
Population: PK analysis set: The sabatolimab and venetoclax pharmacokinetic analysis sets included all participants from the Safety Set who provided at least one evaluable sabatolimab/venetoclax PK concentration. No data is reported as only pre-dose samples were collected
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Trough Serum Concentration (Cmin) Sabatolimab
Description: Concentration of sabatolimab prior to next dosing or after end of treatment by dose level for the safety run-in part (Cohort 1 (400 mg Q4W) and Cohort 2 (800 mg Q4W)).
Time Frame: as for outcome 7
Population: PK analysis set: The sabatolimab pharmacokinetic analysis set included all participants from the Safety Set who provided at least one evaluable sabatolimab PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 5 | 13
ug/ml
  Cycle (C) 1 Day (D) 8: number analyzed (Participants) | 4 | 12
  Cycle (C) 1 Day (D) 8 | 0.0 (0.0) | 0.0 (0.0)
  C2D8: number analyzed (Participants) | 4 | 10
  C2D8 | 23.0 (137.0) | 30.7 (41.7)
  C3D8: number analyzed (Participants) | 1 | 6
  C3D8 | 0.0 (0.0) | 34.4 (72.2)
  C6D8: number analyzed (Participants) | 0 | 3
  C6D8 |  | 68.6 (11.5)
  C9D8: number analyzed (Participants) | 0 | 2
  C9D8 |  | 71.2 (33.8)
  C12D8: number analyzed (Participants) | 0 | 1
  C12D8 |  | 0.0 (0.0)

9. Secondary Outcome: Anti-drug Antibody (ADA) Prevalence at Baseline and ADA Incidence On-treatment by Dose Level
Description: Immunogenicity of sabatolimab prior to sabatolimab exposure and during treatment
Time Frame: as for outcome 7
Population: Immunogenicity (IG) analysis set: included all participants in the Full Analysis Set with a non-missing baseline IG sample or at least one non-missing post-baseline IG sample. A non-missing IG sample was a sample that was analyzed and not ADA-inconclusive.
Measure: Number; unit: Participants
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 4 | 13
Participants
  ADA prevalence at baseline | 0 | 2
  ADA incidence (i.e., ADA positive) on-treatment | 1 | 2
  Treatment-induced ADA-positive | 1 | 1
  Treatment-boosted ADA-positive | 0 | 1

10. Secondary Outcome: Duration of Complete Remission (CR)
Description: Duration of complete remission (CR) is defined as time from first occurrence of CR to relapse from CR, progression or death due to any cause whichever occurs first for the safety run-in part (Cohort 2 (800 mg Q4W)). CR is defined as follows: bone marrow blasts <=5%, hemoglobin level ≥ 10 g/dL, platelets count ≥ 100*10^9/L, neutrophils count ≥ 1.0*10^9/L, absence of blasts in peripheral blood.
  Relapse from complete remission (CR)is when at least 1 of the following criteria is met:
  1. Return to baseline bone marrow blast percentage.
  2. Decrease of ≥ 50% from maximum remission/response levels in neutrophils AND neutrophils <1.0*10^9/L.
  3. Decrease of ≥ 50% from maximum remission/response levels in platelets AND platelets <100*10^9/L.
  4. Decrease from maximum remission/response levels in Hgb concentration by ≥ 1.5g/dL AND Hgb < 10g/dL.
  5. Becoming transfusion dependent
Time Frame: up to approx. 23 months
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) comprises all participants who received at least one dose of study treatment. Analysis is based on participants with CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 1
months | NA [NA to NA] — NA: not enough evens to calculate the median and 95% confidence interval

11. Secondary Outcome: Time to Complete Remission(CR)/Marrow Complete Remission (mCR)
Description: Time to CR/mCR is defined as time from start of treatment to first occurrence of CR or mCR as per investigator assessment for the safety run-in part (Cohort 2 (800 mg Q4W)).
Time Frame: up to approx. 23 months
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) comprises all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 15
months | 2.33 [1.61 to 2.83]

12. Secondary Outcome: Duration of Complete Response (CR)/Marrow Complete Response (mCR)
Description: Duration of CR/mCR is defined as time from first occurrence of CR/mCR to relapse from CR, progression or death due to any cause whichever occurs first for the safety run-in part (Cohort 2 (800 mg Q4W)).
Time Frame: up to approx. 23 months
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) comprises all participants who received at least one dose of study treatment. Analysis is based on participants with CR or mCR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 13
months | 5.60 [4.14 to NA] — NA: with the small sample size and limited follow-up, the survival curve just barely reached the median, so a finite CI upper limit could not be reached.

13. Secondary Outcome: Duration of Response for Participants Who Achieved Hematologic Improvement (HI) or Better
Description: The duration of response was derived for participants treated with sabatolimab at the higher dose who achieved HI or better as per investigator assessment and is defined from the first occurrence of complete response (CR), marrow complete response (mCR), partial response (PR) or hematologic improvement (HI) until relapse, progression or death due to any reason for the safety run-in part (Cohort 2 (800 mg Q4W)).
Time Frame: up to approx. 23 months
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) comprises all participants who received at least one dose of study treatment. Analysis is based on participants with CR, mCR, PR or HI.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 13
months | 5.60 [4.14 to NA] — NA: with the small sample size and limited follow-up, the survival curve just barely reached the median, so a finite CI upper limit could not be reached.

14. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from start of treatment to disease progression (including transformation to acute leukemia per WHO 2016 classification), relapse from CR or death due to any cause, whichever occurs first for the safety run-in part (Cohort 2 (800 mg Q4W)).
Time Frame: up to approx. 23 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 15
months | 6.77 [3.71 to NA] — NA: with the small sample size and limited follow-up, the survival curve just barely reached the median, so a finite CI upper limit could not be reached.

15. Secondary Outcome: Leukemia-Free Survival (LFS)
Description: Time from start of treatment to transformation to acute leukemias per investigator assessment [as defined as ≥ 20% blasts in bone marrow/ peripheral blood (per WHO 2016 classification) or diagnosis of extramedullary acute leukemia or death due to any cause, whichever occurs first for the safety run-in part (Cohort 2 (800 mg Q4W)).
Time Frame: up to approx. 23 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 15
months | 7.59 [4.24 to NA] — NA: with the small sample size and limited follow-up, the survival curve just barely reached the median, so a finite CI upper limit could not be reached.

16. Secondary Outcome: Event-Free Survival (EFS)
Description: Time from start of treatment to lack of reaching CR within the first 6 cycles, relapse from CR or death due to any cause, whichever occurs first for the safety run-in part (Cohort 2 (800 mg Q4W)).
Time Frame: up to approx. 23 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 15
months | 0.03 [NA to NA] — NA: lower and upper limit of 95 Confidence Interval could not be reached because most participants had an EFS event on Day 1 due to treatment failure

17. Secondary Outcome: Overall Survival (OS)
Description: Time from start of treatment to death due to any cause for the safety run-in part (Cohort 2 (800 mg Q4W)).
Time Frame: Date of start of treatment to date of death due to any reason, for up to approx. 23 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 15
months | NA [6.77 to NA] — NA: median and upper limit of 95 Confidence Interval could not be reached because of small sample size and limited survival follow up due to study termination of study

18. Secondary Outcome: Changes in Fatigue (Part 2 - Expansion)
Description: Changes in fatigue as measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue for participants treated with sabatolimab at the higher dose of the expansion part only. Measurements would have been taken via scores from 0 (not at all) to 4 (very much). The higher the score, the better the Quality of Life.
Time Frame: throughout study until progressive disease, death or study discontinuation, approx. 3 years
Population: As expansion phase was not opened, there is no data as nothing was analyzed.
Groups:
- Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 2): Part 2 Expansion: higher dose of sabatolimab in combination with fixed dose of venetoclax and azacitidine.
Arm/Group | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 2)
Number analyzed (Participants) | 0

19. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from start of study treatment (FPFT) up to 30 days after study drug discontinuation, for a maximum duration of approx. 23 months.
  Post-treatment survival follow-up deaths were collected from Day 31 after last dose of study treatment to end of study up to approx. 18 months
  All deaths refer to the sum of on-treatment and post-treatment survival follow-up deaths, up to approx. 23 months
Time Frame: On-treatment deaths: up to approx. 23 months, post-treatment deaths: up to approx 18 months
Population: All enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2)
Number analyzed (Participants) | 5 | 15
Participants
  All deaths | 1 | 6
  On-treatment deaths | 0 | 1
  Post-treatment deaths: number analyzed (Participants) | 5 | 14
  Post-treatment deaths | 1 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 150 days after last dose of study medication (on-treatment), for sabatolimab and 30 days for azactidine & venetoclax up to approx. 23 months. Deaths were collected in the post treatment survival follow up from 31 days after last dose of study medication until the end of the study, up to approx. 18 months. These are not considered AEs
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period.
Groups:
- Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) - On-treatment; Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) - On-treatment: Adverse Events (AEs) during on-treatment period (up to 30 days post-treatment)
- Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) - Post-treatment Survival Follow-up; Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) - Post-treatment Survival Follow-up: Deaths collected in the post- treatment survival follow-up phase (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) - On-treatment | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) - On-treatment | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) - Post-treatment Survival Follow-up | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) - Post-treatment Survival Follow-up
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/15 | 1/5 | 5/14
Serious Adverse Events (participants affected / at risk) | 3/5 | 14/15 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 15/15 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) - On-treatment (N=5) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) - On-treatment (N=15) | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) - Post-treatment Survival Follow-up (N=0) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) - Post-treatment Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | NA | NA
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 5 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | NA | NA
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | NA | NA
Pyrexia (General disorders) | 0 | 1 | NA | NA
Autoinflammatory disease (Immune system disorders) | 0 | 1 | NA | NA
Bacterial sepsis (Infections and infestations) | 1 | 0 | NA | NA
COVID-19 (Infections and infestations) | 0 | 1 | NA | NA
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | NA | NA
Gastroenteritis viral (Infections and infestations) | 0 | 1 | NA | NA
Peritonitis (Infections and infestations) | 0 | 1 | NA | NA
Sepsis (Infections and infestations) | 1 | 1 | NA | NA
Septic shock (Infections and infestations) | 0 | 1 | NA | NA
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Medical observation (Investigations) | 0 | 1 | NA | NA
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) - On-treatment (N=5) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) - On-treatment (N=15) | Sabatolimab (MBG453) 400 mg + AZA + VEN (Part 1 Cohort 1) - Post-treatment Survival Follow-up (N=0) | Sabatolimab (MBG453) 800 mg + AZA + VEN (Part 1 Cohort 2) - Post-treatment Survival Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 7 | NA | NA
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | NA | NA
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 3 | 8 | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 7 | NA | NA
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Sinus bradycardia (Cardiac disorders) | 0 | 1 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | NA | NA
Constipation (Gastrointestinal disorders) | 2 | 4 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | NA | NA
Eructation (Gastrointestinal disorders) | 0 | 1 | NA | NA
Flatulence (Gastrointestinal disorders) | 1 | 0 | NA | NA
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | NA | NA
Nausea (Gastrointestinal disorders) | 1 | 6 | NA | NA
Odynophagia (Gastrointestinal disorders) | 0 | 1 | NA | NA
Stomatitis (Gastrointestinal disorders) | 1 | 3 | NA | NA
Toothache (Gastrointestinal disorders) | 1 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 3 | NA | NA
Asthenia (General disorders) | 1 | 3 | NA | NA
Catheter site inflammation (General disorders) | 0 | 1 | NA | NA
Chills (General disorders) | 0 | 1 | NA | NA
Device related thrombosis (General disorders) | 0 | 1 | NA | NA
Fatigue (General disorders) | 1 | 2 | NA | NA
Hyperthermia (General disorders) | 0 | 1 | NA | NA
Infusion site haematoma (General disorders) | 0 | 1 | NA | NA
Injection site erythema (General disorders) | 0 | 1 | NA | NA
Injection site pain (General disorders) | 0 | 1 | NA | NA
Injection site reaction (General disorders) | 1 | 0 | NA | NA
Oedema peripheral (General disorders) | 0 | 2 | NA | NA
Peripheral swelling (General disorders) | 0 | 1 | NA | NA
Pyrexia (General disorders) | 0 | 2 | NA | NA
Cholestasis (Hepatobiliary disorders) | 1 | 1 | NA | NA
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1 | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | NA | NA
Jaundice (Hepatobiliary disorders) | 0 | 1 | NA | NA
COVID-19 (Infections and infestations) | 0 | 1 | NA | NA
Cellulitis (Infections and infestations) | 0 | 1 | NA | NA
Clostridium bacteraemia (Infections and infestations) | 0 | 1 | NA | NA
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | NA | NA
Oral herpes (Infections and infestations) | 0 | 1 | NA | NA
Sepsis (Infections and infestations) | 0 | 1 | NA | NA
Tooth abscess (Infections and infestations) | 1 | 0 | NA | NA
Vascular device infection (Infections and infestations) | 0 | 1 | NA | NA
Blood bilirubin increased (Investigations) | 0 | 1 | NA | NA
Blood folate decreased (Investigations) | 0 | 1 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | NA | NA
Blood urea increased (Investigations) | 0 | 1 | NA | NA
C-reactive protein increased (Investigations) | 0 | 2 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | NA | NA
Neutrophil count decreased (Investigations) | 1 | 2 | NA | NA
Platelet count decreased (Investigations) | 0 | 3 | NA | NA
Serum ferritin decreased (Investigations) | 0 | 1 | NA | NA
Troponin T increased (Investigations) | 0 | 1 | NA | NA
Weight decreased (Investigations) | 0 | 1 | NA | NA
White blood cell count decreased (Investigations) | 0 | 1 | NA | NA
Cell death (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Gout (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Dizziness (Nervous system disorders) | 0 | 1 | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | NA | NA
Headache (Nervous system disorders) | 0 | 1 | NA | NA
Anxiety (Psychiatric disorders) | 0 | 2 | NA | NA
Confusional state (Psychiatric disorders) | 0 | 1 | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 1 | NA | NA
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | NA | NA
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | NA | NA
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | NA | NA
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Haematoma (Vascular disorders) | 0 | 1 | NA | NA
Hypertension (Vascular disorders) | 0 | 1 | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | NA | NA
Thrombosis (Vascular disorders) | 0 | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04812548/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04812548/SAP_001.pdf